CLINICAL TRIAL: NCT03626480
Title: A Multi-center Longitudinal Cohort Study on Peri-operative Nutrition in Infants With Congenital Heart Disease
Brief Title: Peri-operative Nutrition in Infants With Congenital Heart Disease
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Medical University (Other)
Collaborators: Gansu Provincial Maternal and Child Health Care Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Dalian Children's Hospital (Other)
Responsible Party: Principal Investigator, Yanqin Cui, Director of CICU, Guangzhou Women and Children's Medical Center
Other Study IDs: 2018080101
Record Dates: First submitted 2018-08-01; First posted 2018-08-13 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Congenital Heart Disease
Keywords: Surgery; Nutritional outcome; Infants
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No treatment — No treatment

SUMMARY:
The purpose of our multi-center cohort study is to build a large platform to follow up the peri-operative nutrition of children with congenital heart disease. And data will be collected pre and 1, 3, 6, 12 months post surgery including physical, laboratory, imaging examination and questionnaire. The primary outcome is nutrition status (measured as WAZ, WHZ and HAZ) and secondary outcomes were the biochemical index and quality of life.

DETAILED DESCRIPTION:
Children with congenital heart disease need surgery. However, extracorporeal circulation surgery can lead to systemic inflammatory reaction and ischemia, while reperfusion injury leads to metabolic disorders, with increased metabolism, hyperbolism and reduced anabolism. The redistribution of systemic blood and the ischemic and microcirculatory disorder state of gastrointestinal tract cause damage to the gastrointestinal mucosa and indigestion. Excessive fluid limitation after surgery and positive application of positive inotropic drugs were positively correlated with energy metabolism rate. Additionally, the lack of scientific feeding knowledge and poor eating habits of parents can increase the risk of malnutrition in children. Surgery is the most effective way of treating congenital heart disease. Although the cardiac malformation has been corrected and the heart function has been returned to normal, there are still some children cannot quickly get rid of malnutrition. To our knowledge, postoperative malnutrition affects wound healing in the short term. Long-term malnutrition and lack of calories and protein intake lead to the lack of trace elements, low immune function, easy secondary infection, and affect children's heart, organ function and intellectual development. In conclusion, this group of children with congenital heart disease should draw more extensive attention. And the scientific and reasonable feeding knowledge of infants should be widely carried out, which has far-reaching significance. Therefore, this multi-center cohort study is proposed.

We purposed to carry out a multi-center cohort study, and all infants under 1 year old with congenital heart disease undergone surgery in these hospitals were included. We aimed to follow up a long-term, tracking the nutrition status and motor development. The eligible patients in Guangzhou Women and Children's Medical Center, Shenzhen Children's Hospital, Gansu Provincial Maternity and Child-care Hospital, Zhengzhou Cardiovascular hospital, The Children's Hospital Zhejiang University school of medicine will be included. The baseline data will be collected before surgery, and physical, laboratory and imaging examination will be follow at pre and 1, 3, 6, 12 months post surgery to tracking the change of nutrition status (measured as WAZ, WHZ and HAZ). Questionnaires including emotional and social scales will be assigned pre and post surgery for causal inference and life quality evaluation.

The benefits of our follow up were:

1. patients will be asked to come back to the clinic for periodic review at certain time；
2. specialized people conduct follow up the cohort study；
3. A website system had been established to collect the information of patients:

1) professional CRF forms were unified; 2) the website has quality control features. 3) specialized people are responsible for maintaining the website. 4) the website guarantee the long-distance multi-center communication. 5) the website has a reminder of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All children in the multi-center who met the following criteria:

  1. under 1 years old (including 1 years old);
  2. diagnosed as congenital heart disease and planed to surgery;
  3. parents have basic literacy skills, communication and accessibility
  4. parents are informed consent and volunteered to participate with the approval of the hospital ethics committee,

Exclusion Criteria:

* (1) suspected as chromosomal disease; (2) diagnosis of genetic metabolic diseases; (3) anyway affecting oral feeding (eg. Cleft palate) (4) previous gastrointestinal surgery (eg. Postoperative gastrointestinal fistula)

Ages: 1 Day to 12 Months | Sex: All
Age Groups: Child
Study Population: Infants under 1 years old in the multi-center with congenital heart disease and planed to surgery
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in infants' height and weight | baseline, 1, 3, 6 and 12 months
  Measured as : WAZ (weight-for-age z-score), WHZ (weight-for-height z-score), HAZ (height-for-age z-score). Children's height and weight will be measured pre and 1, 3, 6, 12 months post surgery.

SECONDARY OUTCOMES:
Change of Biomedical index level | baseline, 1, 3, 6 and 12 months
  Infants' Albumin, prealbumin, retinol binding protein (RBP), transferrin (FER) and Amino terminal brain natriuretic peptide precursor (NT-proBNP) will be tested pre and 1, 6 months post surgery.
  Infants' Hemoglobin, microelement, cholesterol, triglyceride and 25-hydroxy vitamin D3 will be tested pre and 3, 12 months post surgery.
Change in ROSS score | baseline, 1, 3, 6 and 12 months
  ROSS score will be evaluated at pre and 1, 3, 6, 12 months post surgery. According to Ross RD, Bollinger RO, Pinsky WW (1992) Grading the severity of congestive heart failure in infants. Pediatr Cardiol 13:72-75. Ross scoring system for heart failure in infants grades the presence and severity of congestive heart failure based on the following variables: amount of formula consumed per feeding, feeding time, history of diaphoresis or tachypnea, growth parameters, respiratory and heart rates, respiratory pattern, perfusion, presence of edema, diastolic filling sounds, and hepatomegaly.
Change in Alberta Infant Motor Scale (AIMS) | baseline, 1, 3, 6 and 12 months
  AIMS score will be evaluated at pre and 1, 3, 6, 12 months post surgery. The AIMS consists of 58 items at 4 different positions: prone (21 items), supine (9 items), sitting (12 items), and standing (16 items). The components tested for each item are based on 3 elements of movement: weight bearing, posture, and antigravity movements. For any item observed by the examiner, 1 point is given, whereas 0 points are given when the item is not observed. The sum of all items observed gives the total raw score, ranging from 0 to 58. The total raw score also can be converted into a percentile rank. High percentile ranks indicate maturity of the infant's gross motor skills.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqin Cui, MPh, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided